CLINICAL TRIAL: NCT04830176
Title: Role of Moringa Dentifirice in the Management of Plaque Induced Gingivitis. A Clinical Crossover Study
Brief Title: Role of Herbal Dentifrices in the Management of Plaque Induced Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Collaborators: A B Shetty Memorial Institute of Dental Science (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: D-F-19-03-04
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Gingiva; Infection; Plaque, Dental
Keywords: miswak; moringa; plaque; gingival bleeding
MeSH Terms: conditions — Infections; Dental Plaque; Plaque, Amyloid; Gingival Hemorrhage | interventions — Dentifrices

STUDY DESIGN:
Intervention Model Description: sample size of 30- First group of 15 subjects recording of plaque and gingival scores were recorded. Patients were given first dentifrice and asked to brush for 72 hours and then asked to report. A washout period of 2 weeks followed. The next round, the subjects were given the second dentifrice and asked to brush for 72 hrs and then after a period of 3days asked to report
Who Masked: Participant, Care Provider
Masking Description: Both the participant and the care provider were masked. They were unaware of the paste they were using as it was marked alphanumerically
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moringa (Active Comparator): First phase of subjects were given dentifrice for brushing
  Interventions: Other: dentifrice
- miswak (Active Comparator): second phase of subjects were given dentifrice for brushing
  Interventions: Other: dentifrice

INTERVENTIONS:
Other: dentifrice — use of dentifrices for brushing

SUMMARY:
The clinical cross over study involves the use of two herbal based dentifirices moringa and miswak and its efficacy in reducing plaque induced gingivitis. The patients selected are provided with details regarding the research format and consent taken.

DETAILED DESCRIPTION:
The clinical cross over study involves use of miswak and moringa dentifrices. The patients selected are 30 in no and are selected based on having gingival inflammation due to plaque accumulation. All other cases related to gingival inflammation along with patients with underlying systemic disease are excluded from the study.

At baseline, plaque and gingival scores are recorded, followed by giving one of the dentifrice to the patient for brushing. The patients are asked to brush twice a day and asked to report after 72 hrs, following which another recording of plaque and gingival scores are recorded.

The patients are then asked to use their own tooth paste for a period of 2 weeks as a wash out period and recalled after this 2 week interval.

The patients are then given the second dentifrice and asked to brush for 72 hrs and then asked to report again for a plaque and gingival score evaluation.

ELIGIBILITY:
Inclusion Criteria:

* subjects having only plaque induced gingival inflammation

Exclusion Criteria:

* Subjects having gingival inflammation related to underling systemic diseases
* Subjects taking medications
* Gingival inflammation related to other causes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
plaque scores | 72 hours
  plaque score recorded using calibrated periodontal probes

SECONDARY OUTCOMES:
Gingival inflammation scores | 72 hours
  Gingival bleeding scores recorded using caliberated periodontal probes

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty Institute of dental sciences, Mangaluru, India

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be shared to other researchers
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data can be accessible in a months time. The data will have unrestricted time frame